CLINICAL TRIAL: NCT06718179
Title: Randomized Comparison of Short Versus 12 Months Prasugrel Plus Aspirin in Patients with Acute Coronary Syndromes Treated with Percutaneous Coronary Intervention and Everolimus-eluting Stents (SORT OUT XII DAPT Duration Trial)
Brief Title: Comparison of Short Versus 12 Months Prasugrel Plus Aspirin in Patients with Acute Coronary Syndromes Treated with Percutaneous Coronary Intervention and Everolimus-eluting Stents
Acronym: SORT OUT DAPT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SORT OUT XII DAPT Duration; 2024-515236-69-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-12; First posted 2024-12-05 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Drug-eluting stent; Dual antiplatelet treatment
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short duration of DAPT (Experimental)
  Interventions: Drug: Short duration of aspirin and prasugrel
- Conventional duration of DAPT (Active Comparator)
  Interventions: Drug: Conventional duration of aspirin and prasugrel

INTERVENTIONS:
Drug: Short duration of aspirin and prasugrel — aspirin 75 mg/day for 1 months plus prasugrel 10 mg/day (5 mg/day) for 1 year, followed by lifelong aspirin 75 mg/day after 1 year
  Arms: Short duration of DAPT
Drug: Conventional duration of aspirin and prasugrel — aspirin 75 mg/day lifelong plus prasugrel 10 mg/day (5 mg/day) for 1 year
  Arms: Conventional duration of DAPT

SUMMARY:
The SORT OUT XII dual antiplatelet treatment (DAPT) duration trial, is a clinical randomized controlled superiority and non-inferiority trial to compare whether prasugrel alone versus prasugrel plus aspirin from month 1 to month 12 after percutaneous coronary intervention with and everolimus-eluting stent in patients with acute coronary syndromes (1) is superior regarding clinically relevant bleeding and (2) non-inferior regarding safety (cardiac death, myocardial infarction, definite stent thrombosis, ischemic stroke or clinically driven target lesion revascularization)

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 years with acute coronary syndromes who are treated with an everolimus-eluting drug-eluting stent can undergo randomization if they can be treated with prasugrel for 12 months.
* Postmenopausal women or use of contraceptive drugs (absence of menstruation in at least 12 consecutive months or continuously usage of contraceptive drugs (a contraceptive implant, an intrauterine device, birth-control pills, transdermal patches, vaginal ring, or depot injection).

Exclusion Criteria:

* Age < 18 years
* Not able to consent to study participating (eg. intubated patients)
* Do not speak Danish
* Life expectancy <1 year
* Allergic to study related treatment
* Non-vitamin K antagonist oral anticoagulants (NOAC) or warfarin treatment
* Contraindication for 12 months prasugrel treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3150 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with clinically relevant bleeding (Effectiveness) | 1 year
  Clinically relevant bleeding is defined a "Bleeding Academic Research Consortium" (BARC) where BARC group 2, 3 and 5 are registered
Number of patients with a composite major adverse cardiovascular or cerebrovascular events (Safety) | 1 year
  Major adverse cardiovascular or cerebrovascular events (MACCE) is defined as a composite of cardiac death, myocardial infarction, definite stent thrombosis, ischemic stroke or clinically driven target lesion revascularization)

SECONDARY OUTCOMES:
Number of patients with clinically relevant bleeding | 1 year
  Clinically relevant bleeding is defined a "Bleeding Academic Research Consortium" (BARC) 2, 3 and 5, where BARC group 2, 3 and 5 are registered
Number of patients with all-cause death | 1 year
  All-cause death is defined as any death
Number of patients with cardiac death | 1 year
  Cardiac death is defined as death resulting from cardiovascular causes: death caused by acute myocardial infarction, death caused by sudden cardiac, including unwitnessed, death, death resulting from heart failure, death caused by cardiovascular procedures. Undetermined cause of death is defined as a death not attributable to any other category because of the absence of any relevant source documents. Such deaths will be classified as cardiovascular for end point determination
Number of patients with myocardial infarction | 1 year
  Myocardial infarction diagnosis follows "The Joint ESC/ACCF/AHA/WHF Task Force on "Third Universal Definition of acute myocardial infarction",which has been adapted by Academy Research Consortium. Acute myocardial infarction not related to other than index lesion is defined as any acute myocardial infarction that is not clearly attributable to a non-target vessel
Number of patients with definite stent thrombosis | 1 year
  Definite stent thrombosis is defined as:
  Angiographic confirmation of stent thrombosis. The presence of a thrombus that originates in the stent or in the segment 5 mm proximal or distal to the stent or in a side branch originating from the stented segment and the presence of at least one of the following criteria:
  Acute onset of ischemic symptoms at rest New electrocardiographic changes suggestive of acute ischemia Typical rise and fall in cardiac biomarkers (refer to definition of spontaneous myocardial infarction) Or Pathological confirmation of stent thrombosis
Number of patients with target lesion revascularization | 1 year
  Target lesion revascularization is defined as a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment including the 5-mm margin proximal and distal to the stent
Number of patients with stroke | 1 year
  Ischemic stroke is defined from the Neurologic Academic Research Consortium (Neuro-ARC):
  Classification on the basis of symptoms and evidence of CNS injury, including overt (acutely symptomatic) CNS injury (Type 1), covert (acutely asymptomatic) CNS injury (Type 2), and neurological dysfunction (acutely symptomatic) without CNS injury (Type 3)
Health-related quality of life | 1 month and 1 year
  Health-related quality of life (HRQoL) will be assessed by the health state classifier EQ-5D
Angina status | 1 month and 1 year
  Angina status is based on the Canadian Cardiovascular Society classification system (SaQ)

CONTACTS AND LOCATIONS:
Overall Officials: Lisette O Jensen, MD, Principal Investigator — Odense University Hospital; Evald H Christiansen, MD, Principal Investigator — Aarhus University Hospital; Ashkan Eftekhari, MD, Principal Investigator — Aalborg University Hospital
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol